CLINICAL TRIAL: NCT03892187
Title: Older Adult Safety in Surgery (OASIS) - Can a Preoperative Self-Reported Functional Status Information Improve Prediction of Cardiac Mobility Related Complications That Threaten Patient Safety In Older Adult Surgical Patients?
Brief Title: Older Adult Safety in Surgery IV (OASIS)
Acronym: OASIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Anesthesia Patient Safety Foundation (Other)
Responsible Party: Principal Investigator, J. Matthias Walz, Chair of Anesthesiology & Perioperative Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H00010380
Record Dates: First submitted 2019-03-21; First posted 2019-03-27 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Frail Elderly Syndrome
Keywords: prehabilitation; perioperative outcomes

STUDY DESIGN:
Intervention Model Description: We will randomize patients in a 1:1 fashion into intervention and control groups using a prespecified table generated by our study statistician. Patients not considered frail
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group (Experimental): Participants are prescribed a walking prescription based on their baseline daily step count. During the interim between the day of consultation until the day of surgery, a study staff member will make weekly calls to each participant. Participants will also log all of their physical activities including the date, activity type, and number of minutes.
  Interventions: Behavioral: Intervention Group
- Control Group (No Intervention): Participants receive usual care prior to surgery. Participants will also log all of their physical activities including the date, activity type, and number of minutes.
- Observation Group (No Intervention): Participants who are not frail will receive usual care prior to surgery and charts will be reviewed for outcomes following surgery.

INTERVENTIONS:
Behavioral: Intervention Group — Walking prescriptions plus weekly coaching calls prior to surgery.
  Arms: Intervention Group

SUMMARY:
Use of remote coaching and walking plan prior to surgery to improve stamina and mobility in frail older adult surgical patients after surgery.

DETAILED DESCRIPTION:
Surgery is a life-saving procedure for patients with cancer and can enhance quality of life for patients with intractable abdominal, urologic, thoracic, or other major disease. Although most patients tolerate the procedure well, frail older adults have as much as a threefold increase in the risk of adverse outcomes after surgery. The proposal will assess the role of a walking intervention in the surgical context over multiple dimensions of physical status-endurance, balance, gait speed, strength, and self-reported function. The investigators will be collecting data on patients who may be undergoing any abdominal, urologic, thoracic, or other major surgery.

The investigators will be introducing a home walking prescription where subjects will self-monitor the amount of walking with use of a fit-bit type wristband pedometer. Via remote coaching and use of the pedometer, the investigators hope to increase the amount of steps over a period of time prior to surgery. A research grade monitor will then be utilized in order to be able to track steps post surgery during the hospital stay. By increasing movement pre and post surgery, the investigators hope to demonstrate that such a program can reduce the incidence of adverse outcomes or improve physical status assessments such as endurance, balance, gait speed, strength, and self-reported function. Patients will be randomized in a 1:1 fashion into intervention and control groups using a prespecified table generated by our study statistician.

Intervention patients will receive a walking prescription and weekly calls from a study staff member. Patients will be given a pedometer to be worn on their wrist, a phone , and a phone charger. Patients will be instructed to synchronize their pedometer to the provided phone once a day. For three days following the baseline visit, patients will be instructed to walk their usual amount. A study staff member will then provide the initial walking prescription based on the participants' baseline performance on the three of baseline walking and will focus the participant on walking at a moderate intensity (level of approximately 3 on the modified Borg Perceived Exertional Scale;14 laminated Borg scales will be distributed to participants).

Participants may walk steps over the course of a day or in one session. The initial walking prescription will also provide instructions to the participant to increase his/her number of steps each week by 10 to 20%.

Study Visits for intervention subjects. Baseline visit (consent)- If agree to participate in the study this group will receive weekly phone calls from a study staff member until the surgery. Following the baseline visit, subjects will also be seen during their preoperative surgical evaluation visit, on the day of their surgery, on approximately the third or fourth day following the surgery or date of discharge if length of stay is less than three days, at approximately 30 days following surgery and a phone call approximately 6 months following the surgery.

Study visits for control frail and control non-frail subjects Baseline visit (consent)- If agree to participate in the study a study staff member will provide general walking advice with typical warnings about when to stop (e.g., chest pain, breathing difficulty, or fall) and will have a follow up phone call approximately 6 months following the surgery. Control subjects will receive no other intervention.

Both groups will be asked to complete a log of their physical activities. Patient data collection will continue for up to one year after the day of surgery.

ELIGIBILITY:
Inclusion criteria:

* Age 60 and older
* Undergoing any abdominal, thoracic, urologic, or other major surgery
* Independently ambulatory
* Patient should be within 3-8 weeks of surgery
* Estimated length of hospital stay after surgery two days or more

Exclusion criteria for screening:

* Non-adults
* Prisoners
* Non-English language speaker for whom short form consent is not available

Exclusion criteria for randomized controlled trial:

* Unstable angina or stable angina with minimal exertion or at rest
* Visual impairment such that walking impairs safety
* Fall within previous three months
* Resting heart rate of more than 120, a systolic blood pressure of more than 180 mm Hg, or a diastolic blood pressure of more than 100 mm Hg
* Patient who does not walk independently (e.g. wheel chair; cane walking is okay)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Distance | 21-45 Days
  Change from baseline 6MWD to 6MWD on day of discharge

SECONDARY OUTCOMES:
Step counts on Post Op days 1 and 2 | 2 days
  Number of steps taken on days one and two post-surgery.
6MWD baseline to presurgical appointment day | 3-6 weeks
  Change from baseline 6MWD to 6MWD on day of presurgical appointment
Baseline to 4 weeks post surgery 6MWD | 7-10 weeks (Baseline can be anywhere between 3 to 6 weeks pre-surgery, therefore 4 weeks post surgery can be anywhere from 7 weeks after baseline to 10 weeks after baseline)
  Change from baseline 6MWD to 6MWD 4 weeks post surgery
Change in The Veterans Rand 12-Item Health Survey (VR12), baseline to 4 wks and 6 months | 7 weeks to 27 weeks
  Change in score on VR12 assessment at baseline as compared to 4 weeks post surgery and 6 months post surgery. The The Veterans Rand 12-Item Health Survey (VR12) is a patient-reported global health measure that is used to assess a patient's overall perspective of their health. Question 1 is on a five point scale, questions 2a and 2b are on a 3 point scale; questions 3 through 5 are on a five point scale, questions 6a -6c are on a six point scale, questions 7 through 9 are on a five point scale. A total score is calculated, with a lower score meaning a more positive perspective of health. We will calculate the total score of the VR12 and then calculate the summary physical component score (PCS) based off of the V12 score, using a published algorithm.16 The algorithm norms PCS to range between 0 and 100, with 50 as a mean, and 10 as the standard deviation for the US population.

CONTACTS AND LOCATIONS:
Overall Officials: Jens M Walz, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Memorial, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Hoque L, Dewolf R, Meyers D, White DK, Mazor KM, Stefan M, Crawford S, Alavi K, Yates J, Maxfield M, Lou F, Uy K, Walz M, Kapoor A. Improving stamina and mobility with preop walking in surgical patients with frailty traits -OASIS IV: randomized clinical trial study protocol. BMC Geriatr. 2020 Oct 7;20(1):394. doi: 10.1186/s12877-020-01799-y. PMID 33028223

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT03892187/Prot_SAP_000.pdf